CLINICAL TRIAL: NCT05745233
Title: The Effect of Intraperitoneal Immune Checkpoint Inhibitor on Malignant Ascites of Patients With Gastric, Pancreatic or Biliary Tract Cancer
Brief Title: Intraperitoneal Immune Checkpoint Inhibitor for Malignant Ascites
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Yuan Bai, Doctor, Division of Hematology and Oncology, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC1-180
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Malignant Ascites
MeSH Terms: interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Checkpoint inhibitor (nivolumab or pembrolizumab) (Experimental): Patients with malignant ascites will received either nivolumab or pembrolizumab intraperitoneally.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nivolumab — Intraperitoneal administration of nivolumab Nivolumab 20 mg in normal saline 100ml will be infused intraperitoneally through a temporary catheter in 10 minutes after paracentesis in a weekly interval.
  Other Names: Opdivo
Drug: Pembrolizumab — Intraperitoneal administration of pembrolizumab Pembrolizumab 20 mg in normal saline 100ml will be infused intraperitoneally through a temporary catheter in 10 minutes after paracentesis in a weekly interval.
  Other Names: Keytruda

SUMMARY:
This projectis aim to evaluate the efficacy of immune checkpoint inhibitor (pembrolizumab or nivolumab) on the malignant ascites of patients with advanced gastric, pancreatic and biliary tract cancers.

DETAILED DESCRIPTION:
Malignant ascites appear when cancer cells metastasize to peritoneal cavity and interfere the circulation of lymph and blood. Patients with malignant ascites suffer from abdominal fullness, abdominal pain, poor intake, decreased nutrition, disability, and eventually inability to further anticancer treatment. Malignant ascites put a heavy burden on patient, their family, society and health care system.

Malignant ascites from cancers of stomach, pancreas and biliary tract are more refractory to intravenous chemotherapy or intraperitoneal chemotherapy than ascites from ovarian or chemo-naïve colorectal cancers because of the inherent nature of chemoresistance. Paracentesis is a treatment with immediate effect but the ascites regrow rapidly and repetitive paracentesis puts patients on the risk of intraabdominal infection. Intraperitoneal infusion of OK-432 can reduce malignant ascites but with intolerable adverse effects of fever, chills, pain, vomiting and septation of ascites which limit the further paracentesis.

Cumulating clinical experience suggests a tolerable safety profile of immune checkpoint inhibitors compared to chemotherapy for patients with malignancy. One theoretical advantage of intraperitoneal administration of immune checkpoint inhibitors is the existence of abundant inflammatory cells, immune cells and mesothelial cells dispersed in the malignant ascites. In addition, both pembrolizumab and nivolumab have been administrated intraperitoneally without obvious toxicities in murine tumor models At China Medical University Hospital, one hundred gastric cancer patients, 50 pancreatic cancer patients and 50 biliary tract cancer patients are registered and treated each year. Among them, more than 20 patients suffer from malignant ascites which will ultimately be managed by repeated paracentesis with increasing frequency. Till now, there is no reported or ongoing clinical trial to investigate the efficacy of intraperitoneal checkpoint inhibitor on the malignant ascites.

ELIGIBILITY:
Inclusion Criteria:

* Patients have cyto-/histologically confirmed malignant ascites from gastric, pancreatic or biliary tract adenocarcinoma
* Patients have malignant ascites more than 1000ml
* Patients have no history of prior intraperitoneal therapy for malignant ascites
* Patients have life expectancy of at least 4 weeks
* Patients have adequate platelet count ≥ 50,000/ul
* Women or men of reproductive potential should agree to use an effective contraceptive method
* All patients must be informed of the investigational nature of this study and must sign written informed consents.

Exclusion Criteria:

* Patients have ascites which is related to causes other than the malignancies
* Patients who are receiving intraperitoneal treatment for their malignant ascites including therapeutic paracentesis
* Patients with active infection
* Patients with bleeding disorders
* Patient with active cardiopulmonary disease or history of ischemic heart disease
* Patients have intolerant abdominal pain
* Patients who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, cirrhosis of the liver, and the rest will be at the discretion of in-charged investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | From the date of registration until the end of treatment, up to 2 years.
  Control of ascites Rate of ascites control = number of patients who have less ascites determinded by five-point method and subjective symptoms / all patients

SECONDARY OUTCOMES:
Adverse effects | From the date of registration until treatment termination, up to 2 years.
  Adverse effect of intraperitoneal immune checkpoint inhibitor Incidence of adverse effect = number of patients who develop a kind of adverse effect / all patients

CONTACTS AND LOCATIONS:
Overall Officials: Li-Yuan Bai, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang ST, Chiu CF, Bai HJ, Bai LY. Intraperitoneal nivolumab in a patient with pancreatic cancer and refractory malignant ascites. Eur J Cancer. 2021 May;148:48-50. doi: 10.1016/j.ejca.2021.01.045. Epub 2021 Mar 15. No abstract available. PMID 33735808
- [Derived] Wang HT, Yu YL, Lo WJ, Lin MC, Chu CL, Chen CY, Wang ST, Chiu CF, Bai EJ, Bai LY. Intraperitoneal nivolumab for malignant ascites in patients with advanced gastrointestinal or pancreaticobiliary tract cancer. Int J Clin Oncol. 2026 Feb;31(2):281-291. doi: 10.1007/s10147-025-02930-y. Epub 2025 Dec 10. PMID 41369826

DOCUMENTS (1):
  • Study Protocol (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT05745233/Prot_000.pdf